CLINICAL TRIAL: NCT05387213
Title: Nurse Practitioner Led Implementation of Team Huddles in Long-Term Care Homes During COVID-19
Brief Title: Nurse Practitioner Led Implementation of Team Huddles in Long-Term Care Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Rehabilitation Institute (Other)
Collaborators: Canadian Foundation for Health Improvement (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government); Centre for Aging and Brain Health Innovation (Other); Walter & Maria Schroeder Institute for Brain Innovation and Recovery (Unknown)
Responsible Party: Principal Investigator, Katherine McGilton, Senior Scientist, Toronto Rehabilitation Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20-6298
Record Dates: First submitted 2022-05-13; First posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Moral Distress; Job Satisfaction; Mental Health; Physical Health; Support
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Huddle attendees (Experimental): Participants in this arm participated in huddles
  Interventions: Behavioral: Team Huddles
- Huddle non-attendees (No Intervention): Participants in this arm did not participate in huddles

INTERVENTIONS:
Behavioral: Team Huddles — Brief multidisciplinary meeting occurring twice a week for staff working at a LTC home led by a Nurse Practitioner. Huddles focused on discussing resident-care and staff-wellbeing.
  Arms: Huddle attendees

SUMMARY:
A pre-experimental design to conduct a process evaluation and to compare the outcomes after implementing team huddles for the intervention and control groups.

DETAILED DESCRIPTION:
Staff working in long-term care (LTC) homes during COVID-19 frequently reported lack of communication, collaboration, and teamwork, all of which are associated with staff dissatisfaction, health concerns, perceived of lack of support and moral distress. The purpose of this study was to introduced regular huddles, led by a Nurse Practitioner, to support LTC staff during COVID-19. The objectives were to evaluate the process of huddle implementation and to examine differences between staff attending and not attending the huddles on outcomes of moral distress, job satisfaction, perceived support from the Nurse Practitioner, and health and mental health. Furthermore, we hypothesize that regular huddles can lead to improvements in resident-centred care and resident outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All staff working at the LTC home
* All residents living in the home between January and December 2021

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Overall morals distress and situations associated with COVID-19 in LTC settings contributing to moral distress were measured in the intervention and control arms using the Moral Distress in Dementia Care Instrument (Iaboni et al., 2021). | 20 weeks
  Moral Distress in Dementia Care is a ten-item checklist, where respondents are asked to rate moral distress associated with each item on a 5-point scale ranging from none (1) to an extremely large amount (5). Higher scores represent more moral distress.
Overall job satisfaction with current role was measured in the intervention and control arms using a single question asking, "How satisfied are you overall with your current job in the LTC home?" (Dolbier et al., 2005) | 20 weeks
  The single-item question was high reliability and validity (Dolbier et al., 2005) and has been used in previous studies in LTC homes (Schwendimann et al., 2016). Respondents rate job satisfaction on a 4-point scale ranging from strongly dissatisfied (1) to strongly satisfied (4), where higher scores indicate more satisfaction.
Overall health was measured in the intervention and control arms using a single question from Statistics Canada (2022) asking, "In general, how would you say your health is?" | 20 weeks
  Respondents rate their health on a 5-point scale ranging from poor (0) to excellent (4), where higher scores indicate better health.
Mental health was measured in the intervention and control arms using a single question from Statistics Canada (2022) asking, "In general, how would you say your mental health is?" | 20 weeks
  Respondents rate their mental health on a 5-point scale ranging from poor (0) to excellent (4), where higher scores indicate better mental health.
Perceived support from the nurse practitioner leading the huddles was measured in the intervention and control arms, assessed using the Supportive Supervisory Scale (McGilton 2010). | 20 weeks
  The 5-item scale asks respondents to rate their perception of support from the nurse practitioner in 5 situations on a 5-point scale ranging from never (0) to always (5), where higher scores indicate more perceived support.

SECONDARY OUTCOMES:
The duration of each huddle in minutes was recorded by the nurse practitioner using the Huddle Observation Tool (HOT) (Edbrooke-Childs et al., 2018) as part of process evaluation. | 15 weeks
  Average and range of huddle duration were measured.
The attendance of different staff categories (i.e. personal support worker, registered practical nurse) at each huddle was recorded by the nurse practitioner using HOT (Edbrooke-Childs et al., 2018) as part of process evaluation. | 15 weeks
  Attendance of categories of staff at huddles was summarized as percentage of total huddles attended.
The frequency of delivery of huddles by the nurse practitioner was self-reported using HOT (Edbrooke-Childs et al., 2018) as part of process evaluation. | 15 weeks
  Data was summarized as total number of huddles delivered and number of huddles delivered per week.
Adherence to huddle structure was self-reported by the nurse practitioner using HOT (Edbrooke-Childs et al., 2018) as part of process evaluation. | 15 weeks
  Data included huddle topic and aim, sharing of a positive event, maintaining a collaborative culture, and creation of a risk management plan and was summarized as number of huddles adhering to the structure.
Depressive symptoms of residents residing on the intervention and control units will be measured with the Depression Rating Scale before and after implementation of huddles. | 1 year
  This is a quality indicator obtained from the Resident Assessment Instrument - Minimum Data Set (RAI-MDS) 2.0. Depression Rating Scale is based on the following items: negative statements (E1a), persistent anger (E1d), expression of unrealistic fears (E1f), repetitive health complaints (E1h), repetitive anxious complaints (E1ii), sad, pained, worried facial expression (E1l), crying, tearfulness (E1m). The score ranges from 0 to 14, where a score of 3 or more may indicate a potential or actual problem with depression.
Aggression of residents residing on the intervention and control units will be measured with the Aggressive Behaviour Scale before and after implementation of huddles. | 1 year
  This is a quality indicator obtained from the RAI-MDS 2.0. Aggressive Behaviour Scale is based on the following items: verbally abusive (E4b), physically abusive (E4c), socially inappropriate/disruptive behaviour (E4d), resists care (E4e). Scores range from 0 to 12, where higher scores indicate higher levels of aggressive behaviour.
The cognitive status of residents on the intervention and control units will be measured with the Cognitive Performance Scale before and after implementation of huddles. | 1 year
  This is a quality indicator obtained from the RAI-MDS 2.0. Cognitive Performance Scale is based on the following items: comatose (B1), short-term memory (B2a), cognition skills for daily decision-making (B4), expressive communication (C4), eating (G1hA). The sores range from 0 to 6, where higher scores indicate more severe cognitive impairment.
Changes in health, end-stage disease, and signs and symptoms of residents on the intervention and control units will be measured using the CHESS scale before and after implementation of huddles. | 1 year
  This is a quality indicator obtained from the RAI-MDS 2.0. CHESS is based on the following items: decline in cognition (B6), decline in ADL (G9), dehydration (J1c), edema (J1g), shortness of breath (J1l), vomiting (J1o), end-stage disease (J5c), weight loss (K3a), leaving food uneaten (K4c). The score ranges from 0 to 5, where higher scores indicate higher levels of medical complexity and are associated with adverse outcomes.
Changes in social engagement of residents on the intervention and control units will be measured with the Index of Social Engagement (ISE) before and after implementation of huddles. | 1 year
  This is a quality indicator obtained from the RAI-MDS 2.0. ISE is based on the following items: at ease interacting with others (F1a), at ease doing planned or structured activities (F1b), at ease doing self-initiated activities (F1c), establishes own goals (F1d), pursues involvement in the life of the facility (F1e), accepts invitations into most group activities (F1f). The scores range from 0-6, where higher scores indicate higher levels of social engagement.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine S McGilton, Principal Investigator — KITE Research Institute - Toronto Rehabilitation Institute
Locations (2):
- Canada (2):
  - Long-Term Care Home, Kitchener, Ontario
  - Long-Term Care Home, Sarnia, Ontario

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers.

REFERENCES:
- [Background] Dolbier CL, Webster JA, McCalister KT, Mallon MW, Steinhardt MA. Reliability and validity of a single-item measure of job satisfaction. Am J Health Promot. 2005 Jan-Feb;19(3):194-8. doi: 10.4278/0890-1171-19.3.194. PMID 15693347
- [Background] Schwendimann R, Dhaini S, Ausserhofer D, Engberg S, Zuniga F. Factors associated with high job satisfaction among care workers in Swiss nursing homes - a cross sectional survey study. BMC Nurs. 2016 Jun 6;15:37. doi: 10.1186/s12912-016-0160-8. eCollection 2016. PMID 27274334
- [Background] McGilton KS. Development and psychometric testing of the Supportive Supervisory Scale. J Nurs Scholarsh. 2010 Jun;42(2):223-32. doi: 10.1111/j.1547-5069.2009.01323.x. PMID 20618606
- [Background] Iaboni A, Quirt H, Engell K, Kirkham J, Stewart S, Grigorovich A, Kontos P, McMurray J, Levy A, Bingham K, Rodrigues K, Astell A, Flint AJ, Maxwell C. Barriers and facilitators to person-centred infection prevention and control: results of a survey about the Dementia Isolation Toolkit. BMC Geriatr. 2022 Jan 25;22(1):74. doi: 10.1186/s12877-022-02759-4. PMID 35078424
- [Background] Edbrooke-Childs J, Hayes J, Sharples E, Gondek D, Stapley E, Sevdalis N, Lachman P, Deighton J. Development of the Huddle Observation Tool for structured case management discussions to improve situation awareness on inpatient clinical wards. BMJ Qual Saf. 2018 May;27(5):365-372. doi: 10.1136/bmjqs-2017-006513. Epub 2017 Sep 19. PMID 28928167
- [Derived] McGilton KS, Krassikova A, Wills A, Bethell J, Boscart V, Escrig-Pinol A, Iaboni A, Vellani S, Maxwell C, Keatings M, Stewart SC, Sidani S. Nurse practitioner led implementation of huddles for staff in long term care homes during the COVID-19 pandemic. BMC Geriatr. 2023 Nov 2;23(1):713. doi: 10.1186/s12877-023-04382-3. PMID 37919676
- See also: Statistics Canada. Canadian Community Health Survey 2022. — http://www.statcan.gc.ca/en/survey/household/3226